CLINICAL TRIAL: NCT03111433
Title: Effect of Coenzyme Q10 on Markers of Endothelial Dysfunction in Pediatric Patients With Type 1 Diabetes Mellitus
Brief Title: Efficacy of Coenzyme q10 in Pediatrics With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Heba ibrahim Mohamed serag, teaching assistant in clinical pharmacy department ,faculty of pharmacy , Ainshams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHCL136
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes mellitus; Coenzyme Q10; endothelial dysfunction; pediatric patients
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — coenzyme Q10; Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental): this group of patients will receive their standard insulin treatment in addition to 100 mg of coenzyme Q10 soft gelatin capsule once daily for three month
  Interventions: Dietary Supplement: Coenzyme Q10; Drug: Insulin
- Group II (Active Comparator): this group of patients will receive their standard insulin treatment only
  Interventions: Drug: Insulin

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Coenzyme Q10 soft gelatin capsule 100mg
  Arms: Group I
Drug: Insulin — multiple dose insulin injection therapy

SUMMARY:
The purpose of this study is to determine wether coenzyme Q10 is effective in reducing markers of endothelial dysfunction in pediatric patients with type 1 diabetes mellitus and aslo to investigate its effect on glycemic control and lipid profile of those patients and its effect on patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age: patients from 8 to 18 years old.
2. Outpatient with at least 1 year history of type 1 diabetes mellitus.
3. Insulin requirement of more than or equal 0.5 U/Kg/day.
4. Approval to participate and give informed consent.

Exclusion Criteria:

1. Presence of systemic disorders such as celiac disease, hypothyroidism or hyperthyroidism.
2. Preexisting cardiovascular disease or hypertension.
3. Chronic kidney disease or chronic liver disease.
4. Significant mental illness.
5. Intake of other antioxidants such as ascorbic acid and α-tocopherol and omega3 supplement within the last 3 months.
6. Intake of coenzyme Q10 within the last 3 months.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2017-03-19 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
change in soluble interacellular adhesion molecule level | three months
  it will be assessed at baseline and after three months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university pediatric's hospital, Cairo, Egypt